CLINICAL TRIAL: NCT06948864
Title: Evaluation of the Role of Preoperative Intravenous Iron in Patients Undergoing Surgery
Brief Title: Evaluate the Outcomes of Ferric Carboxymaltose in Patients With Perioperative Anemia
Status: Completed | Type: Observational
Sponsor: Hospital Universitario Infanta Cristina (Other)
Responsible Party: Principal Investigator, Francisco Javier García Sánchez, PhD. MD. Surgical Prehabilitation Unit Coordinator, Hospital Universitario Infanta Cristina
Other Study IDs: ACT 04/22
Record Dates: First submitted 2025-04-14; First posted 2025-04-29 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Anemia; Anemia (Iron-Loading); Perioperative Bleeding; Infection Prevention; Readmission, Hospital; Surgical Complication; Length of Hospital Stay; Iron Deficiency Anemia Treatment; Prehabilitation
Keywords: infection; anemia; length of stay; prehabilitation
MeSH Terms: conditions — Anemia; Infections | interventions — ferric carboxymaltose

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control (Not surgical prehabilitation): This group received the standard preoperative patient assessment without going through a prehabilitation unit or undergoing any type of intervention. They did not receive this intervention because the surgical prehabilitation consultation had not yet been implemented at the hospital.
- Interventional group (Surgical prehabilitation): This group received standardized care and assessments in a surgical prehabilitation consultation, including preoperative blood tests, correction of conditions such as anemia (including intravenous iron), and the necessary supplementation to optimize the patients.
  Interventions: Drug: Ferric Carboxymaltose (FCM)

INTERVENTIONS:
Drug: Ferric Carboxymaltose (FCM) — Patients in the intervention group underwent surgery from 2020 to end-2022 and were managed according to the surgery prehabilitation protocol. Once the surgeon has included the patient on the SWL, they were evaluated and followed up by the prehabilitation nurse (no more than 72 hours in the case of cancer patients) together with the study internist. The protocol at this preoperative stage consists of a comprehensive biopsychosocial assessment and an analysis of lab and nutritional parameters, which are optimized using targeted treatment. One of the lab parameters analyzed was Hb. Study patients with Hb < 13 g/dL received 500 mg, 1000 mg, 1500 mg or 2000 mg FCM, depending on their levels of Hb, ferritin, transferrin saturation index, and weight. The lab test was repeated immediately before surgery or 30 days after administration of FCM in order to determine whether Hb levels had improved with FCM therapy
  Other Names: infusion
  Groups: Interventional group (Surgical prehabilitation)

SUMMARY:
The prevalence of preoperative anaemia in patients undergoing major surgery is approximately 30%, and is independently associated with higher mortality, a higher rate of postoperative complications, and a greater probability of receiving a transfusion. In a prehabilitation program, the evaluation and correction of anaemia in the preoperative period is essential, as it is a risk factor for transfusions and complications. The main objectives of this study were to analyse the need for blood transfusion, post-surgical complications, hospital length of stay, ICU length of stay, hospital readmissions, and surgical wound infection in patients treated with ferric carboxymaltose (FC) before surgery. A total of 152 patients were included, of whom 96 received FC before the intervention and 56 received no treatment (control group).

DETAILED DESCRIPTION:
It was conducted a prospective pre-post interventional study between 1 January 2019 and 31 December 2022 at Infanta Cristina University Hospital in Parla (Madrid, Spain).

Written informed consent was obtained from each participant. To ensure anonymity and confidentiality, patient data were coded and stored in secure, password-protected databases accessible only to authorized research personnel, in compliance with Spanish legislation (Organic Law 3/2018 and RD 1090/2015).

The data used in the study were anonymous and collected by impartial, unpaid, volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years; on the SWL.
* Hemoglobine <13g/dL.
* Referred for major elective surgery requiring hospital admission (e.g., oncologic resections such as mastectomy, colon resection, nephrectomy, hysterectomy), typically involving general anesthesia and moderate to high morbidity risk, capable of understanding and consenting to the study
* Physically and mentally able to complete assessments

Exclusion Criteria:

* Patients with hypersensitivity to FC, or any of its excipients. • Patients with active bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises patients listed for major oncologic surgeries-such as nephrectomy, mastectomy, colon resection, or hysterectomy-which require general anesthesia and are associated with a high risk of perioperative morbidity and mortality
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Analyze levels of Hemoglobine | From Jan 2019 to Dec 2022
  To analyze the levels of:
  Hemoglobin (Hb) g/dL at three time points:
  Before the administration of intravenous ferric carboxymaltose (FCM), At the time of inclusion on the surgical waiting list, 30 days after surgery. And to compare the incidence of postoperative complications between patients who received FC and those who did not.
Analyze levels of ferritin | From Jan 2019 to Dec 2022
  To analyze the levels of:
  Ferritin (ng/mL)
  at three time points:
  Before the administration of intravenous ferric carboxymaltose (FCM), At the time of inclusion on the surgical waiting list, 30 days after surgery. And to compare the incidence of postoperative complications between patients who received FC and those who did not.
Analyze levels of transferrine | From Jan 2019 to Dec 2022
  To analyze the levels of:
  Transferrin (mg/dL)
  at three time points:
  Before the administration of intravenous ferric carboxymaltose (FCM), At the time of inclusion on the surgical waiting list, 30 days after surgery. And to compare the incidence of postoperative complications between patients who received FC and those who did not.
Analyze levels of transferrine saturation | From Jan 2019 to Dec 2022
  To analyze the levels of:
  Transferrin saturation (%)
  at three time points:
  Before the administration of intravenous ferric carboxymaltose (FCM), At the time of inclusion on the surgical waiting list, 30 days after surgery. And to compare the incidence of postoperative complications between patients who received FC and those who did not.

SECONDARY OUTCOMES:
Compare ferric carboxymaltose vs control (other) | from january 2019 to decembre 2022
  To compare between the groups (ferric carboxymaltose vs. control):
  Hospital length of stay (in days)
Compare ferric carboxymaltose vs control (other) | from january 2019 to decembre 2022
  To compare between the groups (ferric carboxymaltose vs. control):
  ICU admission (yes/no)
Compare ferric carboxymaltose vs control (other) | from january 2019 to decembre 2022
  To compare between the groups (ferric carboxymaltose vs. control):
  ICU length of stay (in days)
Compare ferric carboxymaltose vs control (other) | from january 2019 to decembre 2022
  To compare between the groups (ferric carboxymaltose vs. control):
  Need for hospital readmission (yes/no)
Compare ferric carboxymaltose vs control (other) | from january 2019 to decembre 2022
  To compare between the groups (ferric carboxymaltose vs. control):
  Need for blood transfusion (yes/no)
Compare ferric carboxymaltose vs control (other) | from january 2019 to decembre 2022
  To compare between the groups (ferric carboxymaltose vs. control):
  Surgical wound infection (Yes/no)
Compare ferric carboxymaltose vs control (other) | from january 2019 to decembre 2022
  To compare between the groups (ferric carboxymaltose vs. control):
  Complications (yes/no)
Compare ferric carboxymaltose vs control (other) | from january 2019 to decembre 2022
  To compare between the groups (ferric carboxymaltose vs. control):
  Sepsis (yes/no)
Compare ferric carboxymaltose vs control (other) | from january 2019 to decembre 2022
  To compare between the groups (ferric carboxymaltose vs. control):
  Pleural effusion (yes/no)
Compare ferric carboxymaltose vs control (other) | from january 2019 to decembre 2022
  To compare between the groups (ferric carboxymaltose vs. control):
  Respiratory infection (yes/no)
Compare ferric carboxymaltose vs control (other) | from january 2019 to decembre 2022
  To compare between the groups (ferric carboxymaltose vs. control):
  Abdominal colection (yes/no)
Compare ferric carboxymaltose vs control (other) | from january 2019 to decembre 2022
  To compare between the groups (ferric carboxymaltose vs. control):
  Paralytic ileum (yes/no)
Compare ferric carboxymaltose vs control (other) | from january 2019 to decembre 2022
  To compare between the groups (ferric carboxymaltose vs. control):
  Bleeding (yes/no)
Compare ferric carboxymaltose vs control (other) | from january 2019 to decembre 2022
  To compare between the groups (ferric carboxymaltose vs. control):
  Urinary tract infection (yes/no)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Infanta Cristina, Parla, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
A manuscript for divulgating results.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: End date: May 2025
Access Criteria: Open Access

REFERENCES:
- [Background] Bisbe Vives E. [Treatment of preoperative anemia in major orthopedic surgery]. Rev Esp Anestesiol Reanim. 2015 Jun;62 Suppl 1:52-6. doi: 10.1016/S0034-9356(15)30008-6. Spanish. PMID 26320345
- [Background] Schack A, Berkfors AA, Ekeloef S, Gogenur I, Burcharth J. The Effect of Perioperative Iron Therapy in Acute Major Non-cardiac Surgery on Allogenic Blood Transfusion and Postoperative Haemoglobin Levels: A Systematic Review and Meta-analysis. World J Surg. 2019 Jul;43(7):1677-1691. doi: 10.1007/s00268-019-04971-7. PMID 30824959
- [Background] Munoz M, Aragon S, Ballesteros M, Bisbe-Vives E, Jerico C, Llamas-Sillero P, Meijide-Miguez HM, Rayo-Martin E, Rodriguez-Suarez MJ. Executive summary of the consensus document on the management of perioperative anemia in Spain. Rev Clin Esp (Barc). 2024 Apr;224(4):225-232. doi: 10.1016/j.rceng.2024.02.012. Epub 2024 Feb 27. PMID 38423382
- [Background] Calleja JL, Delgado S, del Val A, Hervas A, Larraona JL, Teran A, Cucala M, Mearin F; Colon Cancer Study Group. Ferric carboxymaltose reduces transfusions and hospital stay in patients with colon cancer and anemia. Int J Colorectal Dis. 2016 Mar;31(3):543-51. doi: 10.1007/s00384-015-2461-x. Epub 2015 Dec 22. PMID 26694926
- [Background] Froessler B, Palm P, Weber I, Hodyl NA, Singh R, Murphy EM. The Important Role for Intravenous Iron in Perioperative Patient Blood Management in Major Abdominal Surgery: A Randomized Controlled Trial. Ann Surg. 2018 Feb;267(2):e39-e40. doi: 10.1097/SLA.0000000000002055. No abstract available. PMID 29300713
- [Background] Garcia Erce JA, Altes A, Lopez Rubio M, Remacha AF; en representacion del Grupo Espanol de Eritropatologia de la Sociedad Espanola de Hematologia y Hemoterapia; Otros componentes del Grupo Espanol de Eritropatologia de la Sociedad Espanola de Hematologia y Hemoterapia. Management of iron deficiency in various clinical conditions and the role of intravenous iron: Recommendations of the Spanish Erythropathology Group of the Spanish Society of Haematology and Haemotherapy. Rev Clin Esp (Barc). 2020 Jan-Feb;220(1):31-42. doi: 10.1016/j.rce.2019.09.004. Epub 2019 Nov 27. English, Spanish. PMID 31783987
- [Background] Laso-Morales M, Jerico C, Gomez-Ramirez S, Castellvi J, Viso L, Roig-Martinez I, Pontes C, Munoz M. Preoperative management of colorectal cancer-induced iron deficiency anemia in clinical practice: data from a large observational cohort. Transfusion. 2017 Dec;57(12):3040-3048. doi: 10.1111/trf.14278. Epub 2017 Aug 21. PMID 28833205
- [Background] Munoz M, Acheson AG, Bisbe E, Butcher A, Gomez-Ramirez S, Khalafallah AA, Kehlet H, Kietaibl S, Liumbruno GM, Meybohm P, Rao Baikady R, Shander A, So-Osman C, Spahn DR, Klein AA. An international consensus statement on the management of postoperative anaemia after major surgical procedures. Anaesthesia. 2018 Nov;73(11):1418-1431. doi: 10.1111/anae.14358. Epub 2018 Jul 31. PMID 30062700
- [Background] Savy M, Edmond K, Fine PE, Hall A, Hennig BJ, Moore SE, Mulholland K, Schaible U, Prentice AM. Landscape analysis of interactions between nutrition and vaccine responses in children. J Nutr. 2009 Nov;139(11):2154S-218S. doi: 10.3945/jn.109.105312. Epub 2009 Sep 30. PMID 19793845
- [Background] Gillis C, Fenton TR, Sajobi TT, Minnella EM, Awasthi R, Loiselle SE, Liberman AS, Stein B, Charlebois P, Carli F. Trimodal prehabilitation for colorectal surgery attenuates post-surgical losses in lean body mass: A pooled analysis of randomized controlled trials. Clin Nutr. 2019 Jun;38(3):1053-1060. doi: 10.1016/j.clnu.2018.06.982. Epub 2018 Jul 9. PMID 30025745
- [Background] Hu WH, Cajas-Monson LC, Eisenstein S, Parry L, Cosman B, Ramamoorthy S. Preoperative malnutrition assessments as predictors of postoperative mortality and morbidity in colorectal cancer: an analysis of ACS-NSQIP. Nutr J. 2015 Sep 7;14:91. doi: 10.1186/s12937-015-0081-5. PMID 26345703
- [Background] Nicholls G, Mehta R, McVeagh K, Egan M. The Effects of Intravenous Iron Infusion on Preoperative Hemoglobin Concentration in Iron Deficiency Anemia: Retrospective Observational Study. Interact J Med Res. 2022 Feb 3;11(1):e31082. doi: 10.2196/31082. PMID 35113024
- [Background] Mudarra-Garcia N, Roque-Rojas F, Izquierdo-Izquierdo V, Garcia-Sanchez FJ. Prehabilitation in Major Surgery: An Evaluation of Cost Savings in a Tertiary Hospital. J Clin Med. 2025 Apr 3;14(7):2460. doi: 10.3390/jcm14072460. PMID 40217909